CLINICAL TRIAL: NCT05357209
Title: Avidhrt Clinical Equivalence of ECG
Brief Title: Avidhrt Clinical Equivalence Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Avidhrt Inc. (Industry)
Collaborators: ASCENSION SACRED HEART (Unknown); Michigan State University (Other); Spring Arbor University (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ACES-01
Record Dates: First submitted 2022-04-27; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Equivalence of ECG Electrode Type Signal Quality for AF and Non AF Users
Keywords: ECG Equivalence

STUDY DESIGN:
Intervention Model Description: This study is divided into two arms. Arm A will contain subjects with diagnosed AF, and arm B will contain all other subjects. This is a prospective, parallel-cohort, non-randomized study using an enriched population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Arm A (Other): Arm A of the Avidhrt study will contain subjects that have been/are diagnosed with AF. Arm A of the study will have the participants complete the Human Factors sub-study in addition to the primary clinical study.
  Interventions: Device: Avidhrt Sense Heart Monitor
- Arm B (Other): Arm B of the Avidhrt study will contain all other subjects (those non diagnosed with AF), and participants will receive the option whether to participate in the Human Factors sub-study.
  Interventions: Device: Avidhrt Sense Heart Monitor

INTERVENTIONS:
Device: Avidhrt Sense Heart Monitor — Use of Avidhrt Sense Heart Monitor review ECG signals.

SUMMARY:
The Avidhrt Clinical Equivalence Study will test and evaluate the equivalency between ECG signals acquired simultaneously using the Avidhrt Sense Lead-1 ECG, and an FDA cleared Lead-12 gel ECG. The Avidhrt Clinical Equivalence Study also includes a sub-study. The Avidhrt Sense Human Factors sub-study will evaluate the usability and efficacy of the user-interface of the Avidhrt Sense device.

DETAILED DESCRIPTION:
This study will test the clinical equivalency of an Avidhrt Sense acquired Lead-I ECG signal and a Lead-I ECG signal obtained from an FDA cleared 12-lead-ECG gel electrode.The Avidhrt Clinical Equivalence study is comprised of study Arm A and Arm B. In Arm A of this study the population is comprised exclusively of subjects with AF, who will be asked to participate in the Clinical Equivalence Study and in the Human Factors Sub-Study. In Arm B of this study the population will consist of all other subjects (no AF), who will be asked to participate in the Clinical Equivalence Study, with the option to enroll and participate in the Human Factors Sub-Study. This is a prospective, parallel-cohort, non-randomized study using an enriched population.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 22 years old at the time of enrollment
* Capable of giving informed consent
* Sufficient manual dexterity to capture an ECG using Avidhrt Sense
* Subjects in the arrhythmia group must have a known history of arrhythmia, and may have an arrhythmia at the time of enrollment based on the screening ECG just before the study recordings are taken.

Exclusion Criteria:

* Cardiac pacemaker or implantable cardioverter-defibrillator
* History of a life-threatening rhythm such as ventricular tachycardia or ventricular fibrillation
* Anti-arrhythmic (rhythm control) medication use (such as amiodarone or flecainide)
* Subjects in the normal controls group should not have any history of arrhythmia and should not be in arrhythmia at the time of enrollment based on the screening ECG
* Subjects with tremors who are unable to stably hold the Avidhrt Sense during a recording without movement

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-05-15 (Estimated); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
Avidhrt Sense ECG equivalency | 12 months